CLINICAL TRIAL: NCT04364282
Title: War of Attrition: Predicting Dropout From Pediatric Weight Management
Brief Title: Stay In Treatment for Pediatric Weight Management
Acronym: SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Boston Children's Hospital (Other); Children's Mercy Hospital Kansas City (Other); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00062191
Record Dates: First submitted 2020-04-21; First posted 2020-04-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Obesity; Attrition; Family Research; Weight Loss
MeSH Terms: conditions — Pediatric Obesity; Tooth Wear; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care team informed (Active Comparator): Participants in this study will be children and their parents taking part in existing pediatric weight-management programs at participating sites. In this group, members of the weight-management care team will be informed of the family's risk profile for attrition.
  Interventions: Other: Care team informed
- Control (Placebo Comparator): Participants in this study will be children and their parents taking part in existing pediatric weight-management programs at participating sites. In this group, members of the weight-management care team will not be informed of the family's risk profile for attrition.
  Interventions: Other: Control

INTERVENTIONS:
Other: Care team informed — Members of the weight-management care team will be informed of the family's risk profile for attrition and may employ additional contacts to enhance chances of retention.
  Arms: Care team informed
Other: Control — Members of the weight-management care team will not be aware of the family's risk profile for attrition.
  Arms: Control

SUMMARY:
Attrition from pediatric weight management programs is unacceptably high, with dropout ranging from 27-73%. This project will utilize a model that predicts dropout from treatment, increasing its power and accuracy through a multi-site observational study. This will result in a powerful tool that will be used to decrease attrition from pediatric weight management, with the potential for widespread dissemination to improve treatment outcomes.

DETAILED DESCRIPTION:
The obesity epidemic is one of the foremost threats to the health of children and adults in the U.S today. Multidisciplinary pediatric weight management programs have been deemed effective, with increased access to these programs strongly advocated. However, the effectiveness of these programs is limited by attrition, with dropout ranging from 27-73%, limiting health benefits to children and inefficiently utilizing already scarce resources. In addition to better understanding the drivers of attrition, being able to predict or forecast dropout holds great potential to improve adherence and outcomes, and modify treatment approaches to best serve the needs of families. Using a model that isolates variables associated with attrition from pediatric weight management to forecast participant dropout, this prospective, longitudinal observational study will collect comprehensive data on child and family-, obesity-, and treatment-related variables In Stage 1, investigators will install an attrition forecasting model, the Outcomes Forecasting System (OFS), in 3 pediatric weight management programs, and build its precision and calibration using a conceptual model of adherence. In Stage 2, we will establish external validation, installing the OFS in a fourth weight management program, and temporal validation through continued use of the OFS within the 3 original sites. The overall goal of this project is to increase the accuracy and power of an attrition prediction model through its installation in weight management programs and to demonstrate its internal, external, and temporal validity. A greater understanding of patient, family, and disease-specific factors that predict dropout from pediatric weight management can be utilized to prevent attrition. By identifying the most pertinent factors driving attrition across weight management sites, new avenues for treatment and prevention will be identified. This project will result in a valuable tool, available for dissemination across a diverse array of clinical programs to improve adherence, decrease costs, and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child is 7-18 years of age
* Participating child has been referred to one of the participating weight management programs, and the family (child-parent dyad) has chosen to participate in said program.
* Participating child is obese (BMI ≥95th percentile for age and sex).
* Participating child provides assent to participation in the research study.
* At least one parent/guardian consents to participate (and consent to child participation).

The parent should be the primary parent accompanying the child to treatment, and the child's primary residence must be with that parent.

- Both members of the parent-child dyad must speak either English or Spanish.

Exclusion Criteria:

* Participating child cannot complete measures and study activities (non-verbal, significant developmental and behavioral challenges).
* Participating child has a chronic illness that impacts weight (i.e. cancer).
* Participating child with a genetic condition (i.e. Prader-Willi) that is associated with excessive weight.
* One member of the parent-child dyad refuses to participate in the study or does not wish to complete 6 months of treatment.
* One member of the parent-child dyad is unable to participate in 6 month follow-up data collection.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1216 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Attrition from weight management | 6 months
  Completion of treatment is defined as completing 6 months of participation in weight-management program (attending the recommended number of visits, and still considered active after 6 months)

SECONDARY OUTCOMES:
Body mass index (BMI) z score | 6 months
  Measured in child only
Percent of the 95th percentile BMI | 6 months
  Measured in child only
Body weight | 6 months
  Measured in parent only
Family Health Habits | 6 months
  The Family Nutrition and Physical Activity (FNPA) Screening tool will be completed by the parent and used to assess eating, activity, and other habits within the family and home environment. No cut points or threshold have been established for determining Healthy vs Unhealthy home environments. Researchers and practitioners should use their own discretion when interpreting scores on the FNPA.
General and psychosocial health (Parent) | 6 months
  The PROMIS-29 Profile 2.0- short forms for adults will be used to assess anxiety, depression, fatigue, pain, physical function, sleep, and ability to participate in social activities.
General and psychosocial health (Child) | 6 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric/Parent Proxy Profile 25- will be used to assess anxiety, depression, fatigue, pain, physical function/mobility, and peer relationships. Child self-report and Parent Proxy Report.
Family function (Parent report) | 6 months
  Parents will complete the Family Assessment Device (FAD), General Functioning subscale (12 item) as a proxy for an overall picture of family function. This self-report questionnaire asks a series of questions on family function and dynamics and parents will be asked to rate their response on a 4-point Likert scale where 1=strongly agree and 4=strongly disagree.
Family function (Child report) | 6 months
  Child will complete the PROMIS Pediatric Family Relationships measure (short form). This self-report questionnaire assesses the child's perception of family interactions. Participants will be asked to respond to questions on a five-point Likert scale ranging from 1 = never to 5 = always.
Household environment (Parent report) | 6 months
  Parents will be asked to complete the Confusion, Hubbub, and Order Scale (CHAOS). The CHAOS measure is a 15-item instrument specifically designed to be administered to parents for assessing chaos in the child's home environment. This 15-item scale is measured using a 4-point Likert scale where 1= very much like your own home and 4=not at all like your own home. Positive items are reverse scored and higher total scores indicate higher levels of chaos and disruption in the home.
Household environment (Child report) | 6 months
  Children will be asked to complete the Children's Report of Parent Behavior Inventory (CRPBI). The CRPBI is a questionnaire that assesses three factors of parenting: acceptance vs. rejection, psychological control vs. autonomy, and firm vs. lax control. Responses are given on a three-point scale, indicating whether an item is like, somewhat like, or not like the parent.
Stress (Parent report) | 6 months
  Parents will complete the Perceived Stress Scale (PSS). The PSS is a 14-item scale that provides a global appraisal of stress by asking respondents to report whether their lives seem to be unpredictable, uncontrollable, or overloaded. Each item is rated on a 5-point scale ranging from never (0) to almost always (4). Positively worded items are reverse scored, and the ratings are summed, with higher scores indicating more perceived stress.
Stress (Child report) | 6 months
  Children will complete the PROMIS Psychological Stress Experience Short Form 4a. This form is designed to capture psychological stress reactions: feeling overwhelmed, perceived lack of control of one's life, and cognitive-perceptual disruption. Items are scored on a 5-point Likert scale where 0=never and 4=always. Higher scores indicate worse psychological stress.
Motivation/self-efficacy | 6 months
  Both parents and children will complete the Importance, Confidence, and Readiness measure. A self-report questionnaire will assess motivation (importance, confidence, and readiness) and participants will be asked to respond to questions on a five-point Likert scale ranging from 1 = not at all to 5 = very.
Health Literacy | 6 months
  Data collectors will administer the Newest Vital Sign (NVS), a health literacy tool, to parents at baseline and follow-up. The NVS is used to measure health literacy and evaluate the impact of low health literacy on a variety of health outcomes. The NVS is based on a nutrition label from an ice cream container. Parents will be given the label and then asked 6 questions about it. The number of correct responses is totaled and higher scores indicate higher levels of health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Skelton, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Children's Mercy Hospital, Kansas City, Missouri
  - Brenner Children's Hospital, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry DC, Rhodes ET, Hampl S, Young CB, Cohen G, Eneli I, Fleischman A, Ip E, Sweeney B, Houle TT, Skelton J. Stay in treatment: Predicting dropout from pediatric weight management study protocol. Contemp Clin Trials Commun. 2021 Jun 9;22:100799. doi: 10.1016/j.conctc.2021.100799. eCollection 2021 Jun. PMID 34169176

DOCUMENTS (1):
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT04364282/ICF_000.pdf